CLINICAL TRIAL: NCT04038671
Title: Activated Carbon Interphase Effect on Surgical Incisions Compared to Two Common Wound Dressings in a Prospective Randomized Control Trial
Brief Title: Activated Carbon Interphase Effect on Surgical Incisions vs.Two Common Wound Dressings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding sponsor decided to move in a different direction and terminated the study before site began patient recruitment.
Sponsor: Brock Liden, DPM (Individual)
Responsible Party: Sponsor-Investigator, Brock Liden, DPM, Principal Invesigator, Liden, Brock, DPM
Organization: Liden, Brock, DPM (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liden20191
Record Dates: First submitted 2019-06-24; First posted 2019-07-31 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Surgical Wound, Healed
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Activated Carbon Dressing (Experimental): A low-adherent, comprised of 100% pure activated carbon and also conforms to body contours to maintain contact with the incision surface. The dressing may be used either dry or moistened with sterilized water over dry or discharging, partial and full thickness wounds.
  Interventions: Device: Activated Carbon Cloth Dressing
- Knitted Cellulose Acetate Mesh (Active Comparator): a non-adhering dressing, comprised of a knitted cellulose acetate mesh impregnated with a specially-formulated petrolatum emulsion.
  Interventions: Device: Knitted Cellulose Acetate Mesh
- Antimicrobial Alginate Dressing with Silver (Active Comparator): a non-adherent antimicrobial alginate dressing with silver
  Interventions: Device: Antimicrobial Alginate Dressing with Silver

INTERVENTIONS:
Device: Activated Carbon Cloth Dressing — Patients will return for weekly follow-up evaluations the first four weeks following surgery and then will return for a final evaluation eight weeks postoperatively. Incision dressings will be changed by the investigator or the investigator's nursing staff at each weekly visit to assess for incision closure and post-surgical wound complications.
  Arms: Activated Carbon Dressing
Device: Knitted Cellulose Acetate Mesh — Patients will return for weekly follow-up evaluations the first four weeks following surgery and then will return for a final evaluation eight weeks postoperatively. Incision dressings will be changed by the investigator or the investigator's nursing staff at each weekly visit to assess for incision closure and post-surgical wound complications.
  Arms: Knitted Cellulose Acetate Mesh
Device: Antimicrobial Alginate Dressing with Silver — Patients will return for weekly follow-up evaluations the first four weeks following surgery and then will return for a final evaluation eight weeks postoperatively. Incision dressings will be changed by the investigator or the investigator's nursing staff at each weekly visit to assess for incision closure and post-surgical wound complications.
  Arms: Antimicrobial Alginate Dressing with Silver

SUMMARY:
This randomized, prospective study evaluates incision closure, post-surgical wound complications, dressing changes, incision/scar appearance, pain associated with dressing changes, and patient satisfaction rates of an activated carbon dressing versus two commercially available wound dressings.

DETAILED DESCRIPTION:
Postoperative incision complications and surgical site infections are risks for patients undergoing surgery. While most surgical incisions heal without complications, postoperative complications, such as erythema, blistering, maceration, scarring, necrosis, and infection, interfere with the normal healing process. Preventing such complications must be a priority, as they may contribute to longer recovery times, as well as increased hospital stays, costs, and morbidity.

Ideally, surgical incision dressings should exhibit the following characteristics:

* promote a moist environment;
* be absorbent, but transparent so fluid accumulation and other complications may be observed;
* be permeable;
* be low adherent to facilitate removal from skin;
* act as a complete barrier to bacteria and water, but not to moisture vapor; and
* feature some flexibility to avoid restricted limb movement and postoperative edema in the incision area [Chen et al; Collins].

However, despite advances in wound dressing designs, there is no consensus regarding the ideal surgical incision dressing. One emerging dressing modality exhibits these key characteristics. This novel activated carbon cloth dressing is low-adherent, comprised of 100% pure activated carbon and also conforms to body contours to maintain contact with the incision surface.

This randomized, prospective clinical trial will compare this activated carbon cloth dressing to two other commercially-available wound dressings, including a non-adherent antimicrobial alginate dressing with silver and a non-adhering knitted cellulose acetate mesh dressing soaked in Povidone-iodine. The primary endpoint is incision coaptation/closure. Secondary endpoints include incision/scar appearance, such as inflammation and edema, odor, pain, patient satisfaction, and number of dressing changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age.
* Patients of both genders and all races.
* Patients undergoing primary, uni- or bilateral operative procedures of the forefoot, midfoot, non-heel posterior foot, ankle, and lower extremity and whose incisions are linear and at least 2 inches in length.
* Patients who are in good general health.
* Patients with no systemic or local active dermatologic disease, such as, but not limited to eczema, psoriasis, skin cancer, scleroderma, or chronic urticaria.
* Patients with vascular disorders must have been treated surgically to be considered for inclusion.
* Patients with diabetes must have ankle brachial index measurements greater than 0.6 to be considered for inclusion.
* Patients who have voluntarily signed the informed consent form, including HIPAA Authorization.

Exclusion Criteria:

* Patients who are younger than 18 years of age.
* Patients undergoing operative procedures involving the heel or whose incisions are non-linear, such as those with curved arches or "S" configurations, and/or are less than 2 inches in length.
* Patients with previous operative procedure around the same area or joint.
* Patients with systemic or local active dermatologic disease, such as but limited to eczema, psoriasis, skin cancer, scleroderma, or chronic urticaria, that might interfere with surgical site evaluation.
* Patients with history of previous local infection.
* Patients with autoimmune conditions.
* Patients with known allergies or topical hypersensitivities to silver or any other components of the study dressings.
* Patients currently taking steroids or other immune modulators know to affect wound healing.
* Patients with vascular disorders that are non-interventional.
* Patients with diabetes who have ankle brachial index measurements less than 0.6 or lower extremities that are non-interventional or by-passable.
* Patients who are considered by the investigator for any reason to be an unsuitable candidate.
* Patients who are unwilling or unable to follow the follow-up evaluation schedules.
* Patients who refuse to voluntarily sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Incision Closure | 4 weeks
  Complete re-epithelialization with no drainage

SECONDARY OUTCOMES:
Post-Surgical Wound Complications | 8 weeks
  Presence of post-surgical wound complication(s) will be monitored
Incision Scar Appearance | 8 weeks
  Patient & Observer Scar Assessment Scale consists of 2 scales; one that the investigator completes and one that the subject completes. The investigator rates vascularization, pigmentation, thickness relief, and pliability on five 10-point numeric scales, with "normal skin" on the left pole and "worst scar imaginable" on the right pole. Patients rate their scar pain & itching, and scar appearance on six 10-point numeric scales, with "no, no complaints" on the left pole and "yes, worst imaginable" on the right pole. Individual items from both scales are summed with higher scores representing poorer scars and lower scores representing scars more closely resembling normal skin. The total score range of the observer scale component is 5 to 50. The total score range of the patient scale component is 6 to 60. The lowest scores, 5 and 6, respectively, reflect normal skin.
Number of Dressing Changes | 8 weeks
  The number of dressing changes will be counted by the investigator or study staff.
Wound odor | 8 weeks
  Patients will rate the odor of their wound using a Visual Analog Scale that consists of 10-cm(100-mm) line with the descriptor "no odor" positioned at the left pole and the descriptor "extremely offensive odor" positioned at the right pole. The lowest score, 0, reflects no wound odor, whereas a score of 10cm/100mm indicates extremely offensive wound odor.
Pain with Dressing Changes | 8 weeks
  Patients will rate their pain associated with the dressing changes using a Visual Analog Scale, as described by Springer BD et al, Am J Orthopedics, 2015. The Visual Analog Scale consists of a 10-cm (100-mm) line with the descriptor "no pain" positioned at the left pole and the descriptor "worst pain imaginable" positioned at the right pole. The lowest score, 0, reflects no pain, whereas a score of 10/100 indicates worst pain imaginable.
Patient Satisfaction | 8 weeks
  Patients will rate their satisfaction of their ability to perform activities of daily living, including ability to perform personal hygiene activities, ability to change clothes, ability to sit comfortably, and ability to sleep comfortably, using a Visual Analog Scales, as described by Springer et al, Am J Orthopedics, 2015. For each of the 4 satisfaction measures, patients will rate their satisfaction on the scale that consists of a 10-cm (100-mm) line, with the descriptor completely unsatisfied" on the left pole and the descriptor "completely satisfied" on the right pole. These 4 satisfaction measures will be averaged for a composite satisfaction measure. An average score of 10/100 would indicate the patient is completely satisfied, whereas an average of 0 would indicate the patient is completely unsatisfied.
Ease of Dressing Changes | 8 weeks
  Investigator or study staff will rate the difficulty of the dressing changes using a Visual Analog Scale that consists of 10-cm(100-mm) line with the descriptor "no difficulty" positioned at the left pole and the descriptor "extreme difficulty" positioned at the right pole. The lowest score, 0, reflects no difficulty with dressing changes, whereas a score of 10cm/100mm indicates most difficulty with the dressing changes.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Circleville Foot & Ankle, LLC, Circleville, Ohio
  - Hocking Valley Community Hospital, Logan, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen KK, Elbuluk AM, Vigdorchik JM, Long WJ, Schwarzkopf R. The effect of wound dressings on infection following total joint arthroplasty. Arthroplast Today. 2017 Jul 3;4(1):125-129. doi: 10.1016/j.artd.2017.03.002. eCollection 2018 Mar. PMID 29560407
- [Background] Collins A. Does the postoperative dressing regime affect wound healing after hip or knee arthroplasty? J Wound Care. 2011 Jan;20(1):11-6. doi: 10.12968/jowc.2011.20.1.11. PMID 21278635
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Kalinski CK, Schnepf M, Laboy D, HernandezL, Nusbaum J, McGrinder B, Comfort C, Alvarez OM. Effectiveness of a Topical Formulation Containing Metronidazole for Wound Odor and Exudate Control. Wounds. 2005;17(4):84-90.
- [Background] Langlois J, Zaoui A, Ozil C, Courpied JP, Anract P, Hamadouche M. Randomized controlled trial of conventional versus modern surgical dressings following primary total hip and knee replacement. Int Orthop. 2015 Jul;39(7):1315-9. doi: 10.1007/s00264-015-2726-6. Epub 2015 Mar 19. PMID 25787680
- [Background] Springer BD, Beaver WB, Griffin WL, Mason JB, Odum SM. Role of Surgical Dressings in Total Joint Arthroplasty: A Randomized Controlled Trial. Am J Orthop (Belle Mead NJ). 2015 Sep;44(9):415-20. PMID 26372751
- [Background] Tustanowski J. Effect of dressing choice on outcomes after hip and knee arthroplasty: a literature review. J Wound Care. 2009 Nov;18(11):449-50, 452, 454, passim. doi: 10.12968/jowc.2009.18.11.44985. PMID 19901873